CLINICAL TRIAL: NCT00396305
Title: Th1 Response to Influenza: Aging and Vaccine Efficacy
Status: Terminated | Phase: Phase 4 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Principal Investigator, Eastern Virginia Medical School
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 05-0070
Record Dates: First submitted 2006-11-02; First posted 2006-11-06 (Estimated); Last update posted 2010-08-27 (Estimated); Status verified 2010-05

CONDITIONS: Influenza
Keywords: Influenza, vaccine, efficacy, elderly
MeSH Terms: conditions — Influenza, Human

ARMS (4):
- Group 2, Control Double Dose (Experimental): 12 elderly and 6 young participants. This group will be vaccinated with a double dose of vaccine without booster on Day 0. These subjects will receive a double-dose of vaccine administered as 2 consecutive injections (2 injections of 0.5 mL) in the same deltoid. The control group for Group 2 is group 1, Cohort 2.
  Interventions: Biological: Trivalent Inactivated Influenza
- Group 3-Control late booster (Experimental): 12 elderly and 6 young participants. This group will be vaccinated with the standard dose of vaccine (0.5 mL) on Day 0 and with a booster dose of vaccine (0.5 mL) on Day 21. The control for Group 3 is Group 1, Cohort 3.
  Interventions: Biological: Trivalent Inactivated Influenza
- Group 1, Control (Active Comparator): 12 elderly and 8 young participants. Group 1 will be further divided into 4 equal cohorts (each containing 3 elderly and 2 young adults). Cohorts 2, 3, and 4 will receive the standard dose of vaccine and placebo (0.5 mL saline) on Day 0, 21, or 7 respectively. Cohort 1 will be vaccinated with the standard dose of vaccine without placebo/vaccine booster.
  Interventions: Drug: Placebo
- Group 4-Control early booster (Experimental): 12 elderly and 6 young participants. This group will be vaccinated with the standard dose of vaccine (0.5 mL) on Day 0 and with a booster dose of vaccine (0.5 mL) on Day 7. The control for Group 4 is Group 1, Cohort 4.
  Interventions: Biological: Trivalent Inactivated Influenza

INTERVENTIONS:
Drug: Placebo — Sterile phosphate buffered saline solution.
  Arms: Group 1, Control
Biological: Trivalent Inactivated Influenza — The trivalent influenza vaccine is a sterile suspension prepared from the allantoic fluids of chicken embryos infected with a specific type of influenza virus. Each 0.5 mL dose of the vaccine contains 15 mcg hemagglutinin (HA) of 3 strains of virus (H1N1, H3N2, and B). The vaccine is a liquid preparation; as such, no diluent is required. It is essentially clear and slightly opalescent in color.
  Arms: Group 2, Control Double Dose; Group 3-Control late booster; Group 4-Control early booster

SUMMARY:
This research study is being done because influenza (flu) affects many people each year throughout the world. The elderly and those with chronic health problems are at greater risk for complications from the flu. The purpose of this research study is to evaluate vaccination strategies in the elderly and others receiving the influenza vaccination in order to increase protection. All subjects will receive the flu vaccine as an injection in the muscle of the upper arm. Participants may receive a booster [an extra dose of vaccine or placebo (inactive substance)] shot. Study participants will include healthy adult volunteers, ages 21-40, 60-89, or 90 years and older. Subjects will be involved in study related procedures for 6 months.

DETAILED DESCRIPTION:
Influenza and pneumonia are the fourth leading cause of death among people aged over 65 years. Influenza also leads as a cause of catastrophic disability, greatly affecting the quality of life of elderly persons. In the United States alone, an estimated 10 billion dollars is spent annually due to the impact of influenza, and this will rise as the population of seniors rapidly expands. Thus, influenza vaccination is recommended for elderly adults. Although it is cost-effective, influenza vaccination only prevents infection in 30 percent-40 percent of those aged over 65, compared to 70 percent-90 percent of those under 65. Reduced influenza vaccine efficacy and greater morbidity and mortality are thought to be largely due to immune senescence, but the underlying mechanism remains poorly understood. A better understanding of immune senescence can ultimately translate into improved effectiveness for a variety of vaccines, including vaccines against bioterrorist attack (such as small pox vaccine), and thereby bring huge advances in disease prevention and billions in cost savings. The commercially available influenza vaccine used in the United States contains inactivated split viral particles of influenza B and two subtypes of influenza A. These vaccines are cost-effective, but far from perfect; up to 61 percent of vaccinated elderly people acquire influenza infection nonetheless. The safety and cost effectiveness of the licensed split influenza virus vaccine is established, reducing researchers' incentive to further improve the vaccine or define the difficult and expensive-to-measure T cell-mediated immunity to it. The ultimate goal of this proposed non-randomized, open-label study is to improve vaccine efficacy in order to reduce morbidity and mortality from influenza and other infectious diseases in elderly people. The primary objective is to examine the safety and immunogenicity of vaccine strategies to enhance the Type 1 Helper Cells (Th1) response by booster at the peak of Influenza specific (IS)-Th1 expansion following first vaccination. The frequency of IS-Th1 and the antibody level on days 7 and 28 will be used as the two main indicators of immunogenicity, although CD8+ T cell response will also be analyzed. The safety profile to be assessed includes immediate adverse events, solicited local and systemic events, and unsolicited adverse events. Seventy-four healthy individuals who are living independently in the communities surrounding the study site will be invited to participate in the trial. Participants between the ages of 21 and 40 years (young cohort) and those 60 years and older (elderly cohort) will be recruited. Participants will be considered active in the trial for 3 months post vaccination. A telephone follow-up visit will be scheduled at 6 months post-vaccination. Four groups of subjects will be recruited: 1 control group (Group 1) and 3 experimental groups (Group 2, Group 3, and Group 4). This study is linked to DMID protocol 05-0125. Protocol 05-0125 contains Part II of this study.

ELIGIBILITY:
Inclusion Criteria:

* Healthy males and females 21 to 40 years of age or between 60 and 89, or 90 years or older at the time of enrollment.
* Subjects must provide written informed consent prior to first study intervention.
* Subject is judged to be healthy on the basis of verbal history and physical examination.
* Subject is able to cooperate with the requirements of the study (must be able to complete the diary cards and will be available for 6 months after enrollment).
* Subject is mentally capable to give consent based on investigator judgment.
* Females of childbearing potential (all women under the age of 40) must agree to use medically approved contraception and must agree to continue using this method for at least three months after enrollment. Females of childbearing potential on hormonal contraception must be stable on hormonal contraception and must agree to use this method of contraception for at least three months after enrollment. Acceptable forms of medically approved contraception include the use of: oral contraceptives, injectable contraceptives (i.e., Depo-Provera), transdermal contraceptives or double barrier method.
* All females 40 years of age and under must have a negative urine pregnancy test prior to any vaccination in this trial. Please note that even those participants that have a history of tubal ligation or hysterectomy or are post menopausal (at least one year of no menses) must still have a negative urine pregnancy test prior to any vaccination in this trial.
* Physical examination must be normal, or abnormal findings must be judged not clinically significant for this patient population by the Physician Investigator.

Exclusion Criteria:

* Had physician-diagnosed influenza at any time during the past two years.
* Received an influenza vaccine 6 months preceding enrollment in the study.
* Received any other vaccine within 30 days before starting this study or plan to receive any vaccine during the 30 days after enrollment.
* Received immunoglobulin therapy or transfusion with blood or blood products within the previous three months.
* Have known chemical dependency liable to compromise immune function (e.g., alcoholism or illegal drug use not including nicotine or caffeine).
* Are allergic to eggs or egg products, contact lens solution, or have ever had a severe reaction to any vaccine.
* Have a history of hypersensitivity (allergy) to thimerosal or formaldehyde.
* Have chronic respiratory illnesses (clinically significant and/or on systemic immunosuppressive medications e.g., asthma, COPD, emphysema).
* Have had symptoms of an active acute respiratory or other active infections or illnesses in the past 72 hours.
* Have a temperature greater than or equal to 100.4 degrees F (38 degrees C) at enrollment.
* Known or suspected diseases of the immune system (i.e., rheumatoid arthritis, lupus erythematosis, lymphoma, HIV, etc.).
* Have active neurologic disorders (i.e., encephalopathy, optic neuritis/neuropathy, partial facial paralysis, and brachial plexus neuropathy).
* Prior history of Guillain-Barré Syndrome.
* Have underlying unstable (require frequent physician office visits, have required a medication change in the past 3 months and/or require frequent medication dose changes) chronic disease such as cardiovascular disease (i.e., uncontrolled hypertension, congestive heart failure, recent heart attack (within past 6 months), cardiomyopathy; diabetes mellitus, liver disease (i.e., hepatitis, cirrhosis), functional or anatomic asplenia, cancer (excluding skin and prostate cancer) or kidney disease.
* Have a history of hematologic malignancy.
* Current treatment with an immunosuppressive medication (i.e., cancer therapeutic agents, corticosteroids, excluding topical and inhaled corticosteroids).
* Pregnant or breastfeeding females or females planning to become pregnant in the next 6 months.
* Have a latex allergy.
* Are participating in another clinical research trial within 30 days of starting this trial or planning to participate in another clinical research trial at any time during this trial.
* Have any condition that would, in the opinion of the investigator, place subject at risk of injury or render subject unable to meet study requirements.

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2006-11; Primary Completion 2007-09 (Actual); Study Completion 2008-01 (Actual)

PRIMARY OUTCOMES:
Immunogenicity: measured by frequency of IS-Th1 and antibody and T cell responses. | Days 7, 28, 56, and 84 following the initial vaccination.
Safety: including rates of serious adverse events (SAEs) and their relationship to vaccination; rates of local or systemic solicited adverse events (AEs) and their categories; and reported unsolicited AEs following vaccination. | Safety evaluation at 4, 14, and 28 days post-vaccination.

CONTACTS AND LOCATIONS:
Locations (1):
- Eastern Virginia Medical School, Norfolk, Virginia, United States